CLINICAL TRIAL: NCT02512263
Title: Assessment of Adherence and Efficiency of a Home-based Training Program on the Muscular Strength, the Endurance and the Quality of Life for Colon Cancer Patients Treated by Chemotherapy
Brief Title: Assessment of Adherence and Efficiency of a Home-based Training Program on Muscular Strength, Endurance and Qol for Colon Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HBTPCoCa
Record Dates: First submitted 2015-07-27; First posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Intervention group (Experimental): They will have to do all the tests and to follow the home-based training program during 9 weeks.
  Interventions: Procedure: Home-based training program
- control group (No Intervention): They will have to do all the tests but not to follow the home-based training program.

INTERVENTIONS:
Procedure: Home-based training program — A home-based training program of 8 exercises to do 5 times a week during 9 weeks
  Arms: Intervention group

SUMMARY:
The purpose is to assess the adherence and the efficiency of a home-based training program on muscular strength, endurance and the quality of life, fatigue, physical activity, anxiety and depression for colon cancer patient treated by chemotherapy.

DETAILED DESCRIPTION:
It's a 9-weeks experimentation with 4 moments (every 3 weeks) to do the tests.

ELIGIBILITY:
Inclusion Criteria:

* Colon cancer patients treated by chemotherapy adjuvant

Exclusion Criteria:

* Patients who have metastasis
* Patients hospitalized during the experimentation
* Patients who have major orthopedic or neurologic problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-10 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Muscular strength measured by Microfet | 15 minutes

SECONDARY OUTCOMES:
Quality of life measured by questionnaire | 3 minutes
Fatigue measured by questionnaire | 3 minutes
Physical activity measured by questionnaire | 3 minutes
Anxiety measured by questionnaire | 3 minutes
Exercise tolerance measured by Six minute walking test | 6 minutes
Depression measured by questionnaire | 3 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium